CLINICAL TRIAL: NCT05588882
Title: A Prospective Randomized Comparison of Topography-Guided LASIK Surgery to Wavefront-Guided LASIK Surgery
Brief Title: Wavefront-guided vs. Topography-guided LASIK
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Stanford University (Other)
Responsible Party: Principal Investigator, Edward E. Manche, Professor of Ophthalmology, Stanford University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 63961
Record Dates: First submitted 2022-10-17; First posted 2022-10-20 (Actual); Last update posted 2024-09-26 (Actual); Status verified 2024-09

CONDITIONS: Myopia
Keywords: wavefront-guided; topography-guided; LASIK
MeSH Terms: conditions — Myopia

STUDY DESIGN:
Intervention Model Description: Participants contribute one eye to each study arm
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Wavefront-guided LASIK (Active Comparator): Wavefront-guided LASIK for myopia and myopic astigmatism
  Interventions: Procedure: Wavefront-guided LASIK
- Topography-guided LASIK (Active Comparator): Topography-guided LASIK for myopia and myopic astigmatism
  Interventions: Procedure: Wavefront-guided

INTERVENTIONS:
Procedure: Wavefront-guided LASIK — Topography-guided utilizes topography mapping to perform the ablation
  Other Names: Topography-guided LASIK
  Arms: Wavefront-guided LASIK
Procedure: Wavefront-guided — Wavefront-guided utilizes aberrometry to perform the ablation
  Arms: Topography-guided LASIK

SUMMARY:
The study is comparing outcomes of wavefront-guided LASIK to topography-guided LASIK in a randomized contralateral fellow eye study in myopic participants.

DETAILED DESCRIPTION:
The purpose of the study is to compare the results of wavefront-guided LASIK surgery to topography-guided LASIK surgery in participants with nearsightedness with or without astigmatism

Three FDA-approved laser devices are being used for the study.

Two excimer lasers are being used for the study. The excimer laser is used to perform the reshaping of the cornea under a LASIK flap to correct nearsightedness, farsightedness and astigmatism. The two lasers being utilized are the Johnson and Johnson Visx CustomVue excimer laser and the Alcon Allegretto laser in the study. Both have received FDA-approval via a PMA pathway.

One femtosecond laser is being used in the study. The femtosecond laser is used to create the LASIK flap during the first part of the LASIK procedure. The Intralase iFS150 femtosecond laser is being used in the study. The femtosecond laser received FDA- approval via a 510k pathway.

All three lasers are being used according to their approved indications.

ELIGIBILITY:
Inclusion criteria.

* Subjects ages 22 to 59with healthy eyes. Nearsightedness between -1.00 diopters and -9.00 diopters.
* Subjects with less than or equal to 3.00 diopters of astigmatism.

Exclusion criteria.

* Subjects under the age of 22 and over the age of 59
* Subjects with excessively thin corneas.
* Subjects with topographic evidence of keratoconus.
* Subjects with ectactic eye disorders.
* Subjects with autoimmune diseases.
* Subjects who are pregnant or nursing.
* Subjects must have similar levels of nearsightedness in each eye. They cannot be more than 1.5 diopter of difference between eyes.
* Subjects with more than 3.00 diopters of astigmatism
* Subjects must have similar levels of astigmatism in each eye. They cannot have more than 1.00 diopters of difference between eyes.

Ages: 22 Years to 59 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Gender Based: Yes
Enrollment: 50 (Actual)
Dates: Start 2022-10-19 (Actual); Primary Completion 2024-09-24 (Actual); Study Completion 2024-09-24 (Actual)

PRIMARY OUTCOMES:
Percentage of eyes achieving uncorrected visual acuity | One year
  Percentage of eyes achieving an uncorrected visual acuity of 20/40, 20/25 ,20/20, 20/16, 20/12.5 and 20/10 at post-operative month twelve

SECONDARY OUTCOMES:
Percentage of eyes with a change in two or more lines of corrected visual acuity | One year
  Percentage of eyes gaining or losing two or more lines of corrected visual acuity Percentage of eyes gaining or losing 2 or more lines of corrected distance visual acuity
Predictability | One year
  Percentage of eyes within +/- 0.50 and +/- 1.00 diopters of the intended corrected
Patient Quality of Vision | One year
  Percentage of patients preferring the eye that underwent either Wavefront-guided or Topography-guided LASIK
Change in corneal epithelial thickness | One year
  We will be measuring the average change in central corneal epithelial thickness from preoperative to post-operative month12 in eyes undergoing Wavefront-guided LASIK and Topography-guided LASIK

CONTACTS AND LOCATIONS:
Overall Officials: Edward E Manche, MD, Principal Investigator — Stanford University
Locations (1):
- Stanford University School of Medicine, Palo Alto, California, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Lu L, Manche E. Prospective, randomized, contralateral eye comparison of wavefront-guided and topography-guided LASIK. J Cataract Refract Surg. 2025 Oct 1;51(10):889-894. doi: 10.1097/j.jcrs.0000000000001703. PMID 40778939